CLINICAL TRIAL: NCT00622635
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter, 3-period, 14-day Crossover Study to Determine the 24 Hour Lung Function Profile of Indacaterol (300 µg Once Daily [od]) in Patients With Moderate-to-severe COPD, Using Open-label Salmeterol (50 µg Twice Daily [Bis in Die, Bid]) as Active Control
Brief Title: A Crossover Study to Determine the 24 Hour Lung Function Profile of Indacaterol in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2340
Record Dates: First submitted 2008-02-04; First posted 2008-02-25 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; indacaterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Indacaterol 300 μg - placebo to indacaterol - salmeterol 50 μg (Experimental): In treatment period 1, patients received indacaterol 300 μg once daily for 14 days via single-dose dry-powder inhaler (SDDPI); in treatment period 2, patients received placebo to indacaterol once daily for 14 days via SDDPI; and in treatment period 3, patients received salmeterol 50 μg twice daily for 14 days via multi-dose dry-powder inhaler (MDDPI). There was a washout period of 14 days between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Salmeterol 50 μg
- Placebo to indacaterol - salmeterol 50 μg - indacaterol 300 μg (Experimental): In treatment period 1, patients received placebo to indacaterol once daily for 14 days via single-dose dry-powder inhaler (SDDPI); in treatment period 2, patients received salmeterol 50 μg twice daily for 14 days via multi-dose dry-powder inhaler (MDDPI); and in treatment period 3, patients received indacaterol 300 μg once daily for 14 days via SDDPI. There was a washout period of 14 days between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Salmeterol 50 μg
- Salmeterol 50 μg - indacaterol 300 μg - placebo to indacaterol (Experimental): In treatment period 1, patients received salmeterol 50 μg twice daily for 14 days via multi-dose dry-powder inhaler (MDDPI); in treatment period 2, patients received indacaterol 300 μg once daily for 14 days via single-dose dry-powder inhaler (SDDPI); and in treatment period 3, patients received placebo to indacaterol once daily for 14 days via SDDPI. There was a washout period of 14 days between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Salmeterol 50 μg
- Placebo to indacaterol - indacaterol 300 μg - salmeterol 50 μg (Experimental): In treatment period 1, patients received placebo to indacaterol once daily for 14 days via single-dose dry-powder inhaler (SDDPI); in treatment period 2, patients received indacaterol 300 μg once daily for 14 days via SDDPI; and in treatment period 3, patients received salmeterol 50 μg twice daily for 14 days via multi-dose dry-powder inhaler (MDDPI). There was a washout period of 14 days between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Salmeterol 50 μg
- Indacaterol 300 μg - salmeterol 50 μg - placebo to indacaterol (Experimental): In treatment period 1, patients received indacaterol 300 μg once daily for 14 days via single-dose dry-powder inhaler (SDDPI); in treatment period 2, patients received salmeterol 50 μg twice daily for 14 days via multi-dose dry-powder inhaler (MDDPI); and in treatment period 3, patients received placebo to indacaterol once daily for 14 days via SDDPI. There was a washout period of 14 days between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Salmeterol 50 μg
- Salmeterol 50 μg - placebo to indacaterol - indacaterol 300 μg (Experimental): In treatment period 1, patients received salmeterol 50 μg twice daily for 14 days via multi-dose dry-powder inhaler (MDDPI); in treatment period 2, patients received placebo to indacaterol once daily for 14 days via single-dose dry-powder inhaler (SDDPI); and in treatment period 3, patients received indacaterol 300 μg once daily for 14 days via SDDPI. There was a washout period of 14 days between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 300 μg; Drug: Placebo to indacaterol; Drug: Salmeterol 50 μg

INTERVENTIONS:
Drug: Indacaterol 300 μg — Indacaterol 300 μg was provided in powder filled capsules with a single-dose dry-powder inhaler (SDDPI).
Drug: Placebo to indacaterol — Placebo to indacaterol was provided in powder filled capsules with a single-dose dry-powder inhaler (SDDPI).
Drug: Salmeterol 50 μg — Salmeterol 50 μg was provided in powder filled capsules with a multi-dose dry-powder inhaler (MDDPI).

SUMMARY:
This study was conducted to provide detailed information on the efficacy of indacaterol in terms of its effect on spirometry assessed forced expiratory volume in 1 second (FEV1) over a 24 hour time period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2006) and:

  1. Smoking history of at least 20 pack-years
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥ 30% of the predicted normal value
  3. Post-bronchodilator FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria:

* Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to screening or during the run-in period
* Patients requiring long-term oxygen therapy (> 15 hours a day) for chronic hypoxemia
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Any patient with active cancer or a history of cancer with less than 5 years disease-free survival time
* Patients with a history of long QT syndrome or whose QTc interval (Bazett's) measured at screening or randomization is prolonged
* Patients who have been vaccinated with live attenuated vaccines within 30 days prior to screening or during the run-in period
* Patients unable to successfully use a dry powder inhaler device or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (7):
  - Novartis Investigator Site, Normal, Illinois
  - Novartis Investigator Site, Shawnee Mission, Kansas
  - Novartis Investigator Site, Lafayette, Louisiana
  - Novartis Investigator Site, Charlotte, North Carolina
  - Novartis Investigator Site, Raleigh, North Carolina
  - Novartis Investigator site, Cincinnati, Ohio
  - Novartis Investigator Site, Spartanburg, South Carolina
- Belgium (3):
  - Novartis Investigator Site, Genk
  - Novartis Investigator Site, Hasselt
  - Novartis Investigator Site, Herentals
- Spain (4):
  - Novartis Investigator Site, Alicante
  - Novartis Investigator site, Alzira
  - Novartis Investigator Site, Madrid
  - Novartis Investigator site, Mataró

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Indacaterol 300 μg - Placebo to Indacaterol - Salmeterol 50 μg | Placebo to Indacaterol - Salmeterol 50 μg - Indacaterol 300 μg | Salmeterol 50 μg - Indacaterol 300 μg - Placebo to Indacaterol | Placebo to Indacaterol - Indacaterol 300 μg - Salmeterol 50 μg | Indacaterol 300 μg - Salmeterol 50 μg - Placebo to Indacaterol | Salmeterol 50 μg - Placebo to Indacaterol - Indacaterol 300 μg
Started | 13 | 11 | 11 | 13 | 10 | 10
Completed | 13 | 10 | 10 | 13 | 9 | 10
Not Completed | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Abnormal test procedure result(s) | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Indacaterol 300 μg - Placebo to Indacaterol - Salmeterol 50 μg | Placebo to Indacaterol - Salmeterol 50 μg - Indacaterol 300 μg | Salmeterol 50 μg - Indacaterol 300 μg - Placebo to Indacaterol | Placebo to Indacaterol - Indacaterol 300 μg - Salmeterol 50 μg | Indacaterol 300 μg - Salmeterol 50 μg - Placebo to Indacaterol | Salmeterol 50 μg - Placebo to Indacaterol - Indacaterol 300 μg
Started | 13 | 10 | 10 | 13 | 9 | 10
Completed | 12 | 10 | 10 | 13 | 9 | 10
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Indacaterol 300 μg - Placebo to Indacaterol - Salmeterol 50 μg | Placebo to Indacaterol - Salmeterol 50 μg - Indacaterol 300 μg | Salmeterol 50 μg - Indacaterol 300 μg - Placebo to Indacaterol | Placebo to Indacaterol - Indacaterol 300 μg - Salmeterol 50 μg | Indacaterol 300 μg - Salmeterol 50 μg - Placebo to Indacaterol | Salmeterol 50 μg - Placebo to Indacaterol - Indacaterol 300 μg
Started | 12 | 10 | 10 | 13 | 9 | 10
Completed | 12 | 10 | 10 | 10 | 9 | 10
Not Completed | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The entire study population included all 6 treatment groups who received indacaterol 300 µg once daily, placebo to indacaterol once daily, and salmeterol 50 µg twice daily via a single-dose (indacaterol and placebo to indacaterol) or multi-dose (salmeterol) dry-powder inhaler in 6 different sequences. Patients received each treatment for 14 days with a 14 day washout between each treatment period. Indacaterol and placebo to indacaterol were administered double-blind; salmeterol was administered open-label. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 65.6 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of Each Treatment Period (Day 15)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of each treatment period. The analysis included baseline FEV1, defined as the average of the FEV1 values measured at 50 and 15 minutes prior to the first study drug administration in that period, as a covariate.
Time Frame: After 14 days
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol 300 μg: Indacaterol 300 µg was inhaled once daily for 14 days using a single-dose dry-powder inhaler (SDDPI) device. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Placebo to Indacaterol: Placebo to indacaterol was inhaled once daily for 14 days using a single-dose dry-powder inhaler (SDDPI) device. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Salmeterol 50 μg: Salmeterol 50 µg was inhaled twice daily for 14 days using a multi-dose dry-powder inhaler (MDDPI) device. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 61 | 61 | 59
Liters | 1.46 (0.027) | 1.26 (0.027) | 1.37 (0.027)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 5 Minutes Post-dose at the End of Each Treatment Period (Day 14)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The analysis included baseline FEV1, defined as the average of the FEV1 values measured at 50 and 15 minutes prior to the first study drug administration in that period, as a covariate.
Time Frame: 5 minutes post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 64 | 60
Liters | 1.44 (0.022) | 1.24 (0.022) | 1.36 (0.022)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 15 Minutes Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 15 minutes post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 64 | 64 | 59
Liters | 1.47 (0.023) | 1.27 (0.023) | 1.41 (0.024)

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 30 Minutes Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 30 minutes post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 64 | 64 | 60
Liters | 1.49 (0.023) | 1.26 (0.023) | 1.42 (0.024)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 1 Hour Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 1 hour post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 64 | 64 | 60
Liters | 1.49 (0.023) | 1.26 (0.023) | 1.42 (0.023)

6. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 2 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 2 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 64 | 62 | 60
Liters | 1.50 (0.024) | 1.27 (0.024) | 1.44 (0.025)

7. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 3 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 3 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 64 | 61 | 60
Liters | 1.51 (0.023) | 1.29 (0.024) | 1.45 (0.024)

8. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 4 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 4 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 60 | 59
Liters | 1.49 (0.023) | 1.29 (0.023) | 1.44 (0.023)

9. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 5 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 5 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 59 | 59
Liters | 1.49 (0.025) | 1.26 (0.026) | 1.45 (0.026)

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 6 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 6 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 57 | 59
Liters | 1.48 (0.025) | 1.29 (0.026) | 1.42 (0.025)

11. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 8 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 8 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 56 | 59
Liters | 1.44 (0.025) | 1.27 (0.026) | 1.40 (0.026)

12. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 10 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 10 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 56 | 58
Liters | 1.43 (0.024) | 1.25 (0.026) | 1.36 (0.025)

13. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 11 Hours 10 Minutes Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 11 hours 10 minutes post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 55 | 57
Liters | 1.45 (0.025) | 1.25 (0.027) | 1.35 (0.027)

14. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 11 Hours 45 Minutes Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 11 hours 45 minutes post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 63 | 54 | 57
Liters | 1.46 (0.026) | 1.24 (0.028) | 1.35 (0.027)

15. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 14 Hours Post-dose at the End of Each Treatment Period (Day 14)
Description: as for outcome 2
Time Frame: 14 hours post-dose at the end of each treatment period (Day 14)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 61 | 55 | 58
Liters | 1.45 (0.026) | 1.24 (0.027) | 1.39 (0.026)

16. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 20 Hours 10 Minutes Post-dose at the End of Each Treatment Period (Day 15)
Description: as for outcome 2
Time Frame: 20 hours 10 minutes post-dose at the end of each treatment period (Day 15)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 60 | 57 | 61
Liters | 1.36 (0.027) | 1.17 (0.028) | 1.31 (0.027)

17. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 20 Hours 45 Minutes Post-dose at the End of Each Treatment Period (Day 15)
Description: as for outcome 2
Time Frame: 20 hours 45 minutes post-dose at the end of each treatment period (Day 15)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 62 | 59 | 59
Liters | 1.40 (0.025) | 1.19 (0.026) | 1.35 (0.026)

18. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 22 Hours Post-dose at the End of Each Treatment Period (Day 15)
Description: as for outcome 2
Time Frame: 22 hours post-dose at the end of each treatment period (Day 15)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 62 | 60 | 59
Liters | 1.43 (0.026) | 1.25 (0.026) | 1.38 (0.026)

19. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 23 Hours 10 Minutes Post-dose at the End of Each Treatment Period (Day 15)
Description: as for outcome 2
Time Frame: 23 hours 10 minutes post-dose at the end of each treatment period (Day 15)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 61 | 61 | 59
Liters | 1.48 (0.030) | 1.24 (0.030) | 1.37 (0.031)

20. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 23 Hours 45 Minutes Post-dose at the End of Each Treatment Period (Day 15)
Description: as for outcome 2
Time Frame: 23 hours 45 minutes post-dose at the end of each treatment period (Day 15)
Population: Modified intent-to-treat (modified ITT) population: All randomized patients who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 300 μg | Placebo to Indacaterol | Salmeterol 50 μg
Number analyzed (Participants) | 61 | 61 | 59
Liters | 1.45 (0.026) | 1.28 (0.026) | 1.38 (0.026)

ADVERSE EVENTS:
Arm/Group | Indacaterol 300 μg | Salmeterol 50 μg | Placebo to Indacaterol
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/65 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/65 | 4/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=66) | Salmeterol 50 μg (N=65) | Placebo to Indacaterol (N=66)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 300 μg (N=66) | Salmeterol 50 μg (N=65) | Placebo to Indacaterol (N=66)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.